CLINICAL TRIAL: NCT05746091
Title: Arthroscopic Partial Trapeziectomy With Hematoma Distraction in Basal Thumb Arthritis
Brief Title: Arthroscopic Partial Trapezictomy With Hematoma Distraction in Basal Thumb Arthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Abbas Mahmoud, principal investigator, Al-Azhar University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APTBA
Record Dates: First submitted 2023-02-17; First posted 2023-02-27 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Orthopedic Disorder
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arthroscopic partial Trapezictomy With Hematoma Distraction (Experimental)
  Interventions: Procedure: wrist arthroscopy

INTERVENTIONS:
Procedure: wrist arthroscopy — Arthroscopic Partial Trapeziectomy with Hematoma Distraction in Basal Thumb Arthritis

SUMMARY:
The basal joint, also referred to as the carpometacarpal (CMC) joint, of the thumb is one of the joints most commonly affected by arthritis. CMC joint arthritis can lead to decreased grip and pinch strength and impairment of activities of daily living

DETAILED DESCRIPTION:
The thumb CMC joint has been reported as the most painful joint when compared to other hand joints affected by OA. It is therefore no surprise that this is a common chief complaint of patients and has a significant effect on work and life satisfaction Patients often present with complaints of pain localized to the base of the thumb that is exacerbated when performing tasks such as opening a jar, turning a car key, and turning door Knob, this pain may be reproduced by resisted pinch and grip .

On physical examination, patients will have point tenderness at the thumb basal joint with swelling and crepitus when the basal joint is compressed - a positive grind test and a positive "hump" sign from dorsal CMC dislocation subluxation .

ELIGIBILITY:
Inclusion Criteria:

* Age: adult patient > 20years.
* Gender: Males & Females.
* Symptomtic patient.
* Failed conservative treatment of 6 months duration
* Eaton stage II, III and IV of base thumb arthritis

Exclusion Criteria:

* Patient presenting with flexor carpi radialis rupture
* Previous Zancolli arthroplasty
* Associated comorbidity as: RA,DM with joint destruction
* Infection
* Poor Skin Condition
* Active Pateint With High Joint Demand

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2023-12-30 (Actual); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-05 (Estimated)

PRIMARY OUTCOMES:
DASH score | 1 year
  score for pinch grip

CONTACTS AND LOCATIONS:
Locations (1):
- Alazhar, Asyut, Egypt